CLINICAL TRIAL: NCT03093870
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of Varlitinib Plus Capecitabine Versus Placebo Plus Capecitabine in Patients With Advanced or Metastatic Biliary Tract Cancer as Second Line Systemic Therapy
Brief Title: Varlitinib in Combination With Capecitabine for Advanced or Metastatic Biliary Tract Cancer
Acronym: TreeTopp
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Collaborators: bioRASI, LLC (Industry); CMIC Co, Ltd. Japan (Industry); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASLAN001-009
Record Dates: First submitted 2017-03-16; First posted 2017-03-28 (Actual); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-06

CONDITIONS: Biliary Tract Cancer
Keywords: Neoplasms; Biliary Tract Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms; Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — ARRY-334543; Capecitabine

STUDY DESIGN:
Intervention Model Description: Treatment: protocol designed to evaluate one or more interventions for treating a disease, syndrome or condition
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Varlitinib and Capecitabine (Experimental)
  Interventions: Drug: Varlitinib; Drug: Capecitabine
- Placebo and Capecitabine (Placebo Comparator)
  Interventions: Drug: Capecitabine; Drug: Placebo (for Varlitinib)

INTERVENTIONS:
Drug: Varlitinib — Varlitinib:300mg, oral tablets, twice daily. Number of cycles: until disease progression, unacceptable toxicity, withdrawal of consent, or death.
  Other Names: ASLAN001; ARRY-334543; QBT01
  Arms: Varlitinib and Capecitabine
Drug: Capecitabine — 1000mg/m2, oral tablets, twice daily for 2 weeks followed by a 1-week rest period in 3-week cycles. Number of cycles: until disease progression, unacceptable toxicity, withdrawal of consent, or death.
Drug: Placebo (for Varlitinib) — oral tablets, twice daily. Number of cycles: until disease progression, unacceptable toxicity, withdrawal of consent, or death
  Arms: Placebo and Capecitabine

SUMMARY:
This protocol for Varlitinib is developed for the treatment of Biliary Tract Cancer. Varlitinib (also known as ASLAN001) is a small-molecule, adenosine triphosphate competitive inhibitor of the tyrosine kinases - epidermal growth factor receptor (EGFR), human epidermal growth factor receptor (HER)2, and HER4. Varlitinib may be beneficial to subjects with cancer by simultaneous inhibition of these receptors. The purpose of this study is to determine the safety and efficacy of Varlitinib in combination with capecitabine for the treatment of Biliary Tract Cancer. Treatment groups are Varlitinib+capecitabine and Placebo + capecitabine

DETAILED DESCRIPTION:
Part 1 of study(Phase 2) is planned to have 120 patients and anticipated completion on July 2019. Recruitment completed.

Part 2 of study(Phase 3) is planned to have 350 patients and anticipated completion on Dec 2022. Not yet recruiting.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for the study if they:

1. Are of or older than the legal age in the respective countries at the time when written informed consent is obtained
2. Have histologically or cytologically confirmed advanced (unresectable) or metastatic biliary tract cancer, including intrahepatic or extrahepatic cholangiocarcinoma (CCA), gallbladder cancer and carcinoma of Ampulla of Vater. This includes clinical diagnosis of biliary tract cancer with histological confirmation of adenocarcinoma.
3. Have received and failed one and only one prior line of systemic treatment for advanced or metastatic disease with radiologic evidence of disease progression. This prior line of systemic treatment must also contain gemcitabine
4. Have received at least 6 doses of gemcitabine containing treatment in first line (Adjuvant therapy is not regarded as 1st line therapy)
5. Have radiographically measurable disease based on Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 as assessed by Independent Central Review (ICR) (For Part 1)
6. Have no evidence of biliary duct obstruction, unless obstruction is controlled by local treatment or, in whom the biliary tree can be decompressed by endoscopic or percutaneous stenting with subsequent reduction in bilirubin to below or equal to 1.5 × upper level of normal (ULN)
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Are able to understand and willing to sign the informed consent form
9. Have adequate organ and hematological function:

   1. Hematological function, as follows:

      * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
      * Platelet count ≥ 100 × 109/L
   2. Renal functions, as follows:

      • Estimated glomerular filtration rate or creatinine clearance > 50 mL/min/1.73m2
   3. Hepatic function, as follows:

      * Albumin ≥ 3 g/dL
      * Total bilirubin ≤ 1.5 × ULN
      * Aspartate aminotransferase and alanine aminotransferase ≤ 5 × ULN

Exclusion Criteria:

Subjects will be ineligible for the study if they:

1. Are currently on or have received anti-cancer therapy within the past 3 weeks before receiving the first dose of study medication
2. Are currently on or have received radiation or local treatment within the past 3 weeks for the target lesion(s) before receiving the first dose of study medication
3. Have evidence of multiple (≥ 2) peritoneal metastases or ascites at baseline as assessed by ICR (For Part 1). (Ascites which can be attributed by non-malignant causes is not excluded. Minimal ascites, which does not require paracentesis is permitted.)
4. Have had major surgical procedures within 14 days prior to first dose of study medication
5. Have a known metastatic brain lesion(s), including asymptomatic and well controlled lesion(s)
6. Have malabsorption syndrome, diseases significantly affecting gastrointestinal function, resection of the stomach or small bowel, or difficulty in swallowing and retaining oral medications which in the opinion of the Investigator could jeopardize the validity of the study results
7. Have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, diabetes, hypertension, or psychiatric illness/social situations that would limit compliance with study requirements
8. Have any history of other malignancy unless in remission for more than 1 year (non-melanoma skin carcinoma and carcinoma-in-site of uterine cervix treated with curative intent is not exclusionary)
9. Are female patients who are pregnant or breast feeding
10. Have been previously treated with varlitinib or have been previously treated with capecitabine as first line therapy for advanced or metastatic disease. For patients who have previously received capecitabine as a radiosensitizer or as part of their adjuvant therapy and their disease has relapsed for more than 6 months after their last dose of capecitabine adjuvant therapy, their capecitabine therapy will not be considered as a line of systemic chemotherapy for metastatic/advanced disease, and thus they can participate in the study
11. Have received any investigational drug (or have used an investigational device) within the last 14 days before receiving the first dose of study medication
12. Have unresolved or unstable serious toxicity (≥ common terminology criteria for adverse events [CTCAE] 4.03 Grade 2), with the exception of anemia, asthenia, and alopecia, from prior administration of another investigational drug and/or prior cancer treatment
13. Have a known positive test for human immunodeficiency virus, hepatitis C (treatment naïve or after treatment without sustained virologic response), or hepatitis B infection with hepatitis B virus deoxyribonucleic acid exceeding 2000 IU/mL
14. Have a known history of drug addiction within last 1 year which, in the opinion of the Investigator, could increase the risk of non-compliance to investigational product
15. Need continuous treatment with proton pump inhibitors during the study period
16. Have a history of (non-infectious) pneumonitis that required steroids or current pneumonitis, or have a history of interstitial lung disease or current interstitial lung disease
17. Have any history or presence of clinically significant cardiovascular, respiratory, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease or any other condition which in the opinion of the Investigator could jeopardize the safety of the patient or the validity of the study results
18. Have a baseline corrected QT interval (Fridericia's formula) (QTcF) > 450 ms or patients with known long QT syndrome; torsade de pointes; symptomatic ventricular tachycardia; an unstable cardiac syndrome in the past 3 months before screening visit; > class 2 New York Heart Association heart failure; or > class 2 angina pectoris; or receiving quinidine, procainamide, disopyramide, amiodarone, dronedarone, arsenic, dofetilide, sotalol, or methadone. Please also see prohibited medication/therapy (Section 5.4.10.1)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2020-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (11):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Karmanos Cancer Institute/Wayne State University, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - CCCN, Las Vegas, Nevada
  - Ruttenberg Cancer Center, Mount Sinai Hospital, New York, New York
  - Levine Cancer Institute, Carolinas Healthcare System, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology, P.A., Dallas, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
- There are 5 sites in different cities in Australia, Camperdown, Australia
- There are 6 sites in different cities in China, Nanjing, Nanjing, China
- There are 2 sites in Hong Kong, Hong Kong, Hong Kong
- There are 2 sites in Hungary, Budapest, Hungary
- There are 7 sites in different cities in Japan, Chiba, Japan
- There are 2 sites in different cities in Poland, Otwock, Poland
- There are 2 sites in Singapore., Singapore, Singapore
- There are 15 sites in different cities in South Korea, Seoul, South Korea
- There are 5 sites in different cities in Spain, Barcelona, Spain
- There are 5 sites in different cities in Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Period 1: Safety lead-in, N=24. Period 2: Part 1, N=127
Pre-assignment Details: Period 1: Safety lead-in phase had only 1 arm (Varlitinib and Capecitabine). Period 2: Part 1 phase had 2 arms (Varlitinib and Capecitabine vs Placebo and Capecitabine)
Groups:
- Varlitinib and Capecitabine - Safety Lead-In; Varlitinib and Capecitabine - Part 1: Varlitinib: Varlitinib:300mg, oral tablets, twice daily. Number of cycles: until disease progression, unacceptable toxicity, withdrawal of consent, or death.
  Capecitabine: 1000mg/m2, oral tablets, twice daily for 2 weeks followed by a 1-week rest period in 3-week cycles. Number of cycles: until disease progression, unacceptable toxicity, withdrawal of consent, or death.
- Placebo and Capecitabine - Part 1: Placebo (for Varlitinib): oral tablets, twice daily. Number of cycles: until disease progression, unacceptable toxicity, withdrawal of consent, or death.
  Capecitabine: 1000mg/m2, oral tablets, twice daily for 2 weeks followed by a 1-week rest period in 3-week cycles. Number of cycles: until disease progression, unacceptable toxicity, withdrawal of consent, or death.
Period: Overall Study
Arm/Group | Varlitinib and Capecitabine - Safety Lead-In | Varlitinib and Capecitabine - Part 1 | Placebo and Capecitabine - Part 1
Started | 24 | 64 | 63
Completed | 0 | 23 | 22
Not Completed | 24 | 41 | 41
Not completed — Withdrawal by Subject | 2 | 6 | 5
Not completed — Death | 1 | 35 | 35
Not completed — Radiographic disease progression | 10 | 0 | 0
Not completed — Clinical disease progression | 1 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Adverse Event | 7 | 0 | 0
Not completed — Patient withdrew from treatment voluntarily due to intermittent constipation and anorexia | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varlitinib and Capecitabine - Safety Lead-In | Varlitinib and Capecitabine - Part 1 | Placebo and Capecitabine - Part 1 | Total
Number analyzed (Participants) | 24 | 64 | 63 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The study consists of Safety Lead-In (24 patients in Varlitinib + Capecitabine group) and Part 1 (64 patients in Varlitinib + Capecitabine group, 63 patients in Placebo + Capecitabine group)
  years
    Safety Lead-In: number analyzed (Participants) | 24 | 0 | 0 | 24
    Safety Lead-In | 58.5 (9.68) |  |  | 58.5 (9.68)
    Part 1: number analyzed (Participants) | 0 | 64 | 63 | 127
    Part 1 |  | 61.6 (10.39) | 62.7 (11.19) | 62.1 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The study consists of Safety Lead-In (24 patients in Varlitinib + Capecitabine group) and Part 1 (64 patients in Varlitinib + Capecitabine group, 63 patients in Placebo + Capecitabine group)
  Participants
    Safety Lead-In: number analyzed (Participants) | 24 | 0 | 0 | 24
    Safety Lead-In: Female | 13 |  |  | 13
    Safety Lead-In: Male | 11 |  |  | 11
    Part 1: number analyzed (Participants) | 0 | 64 | 63 | 127
    Part 1: Female |  | 20 | 30 | 50
    Part 1: Male |  | 44 | 33 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Overall Study: Hispanic or Latino | 4 | 1 | 1 | 6
  Overall Study: Not Hispanic or Latino | 20 | 63 | 62 | 145
  Overall Study: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Overall Study: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Overall Study: Asian | 9 | 42 | 47 | 98
  Overall Study: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Overall Study: Black or African American | 0 | 1 | 0 | 1
  Overall Study: White | 12 | 21 | 16 | 49
  Overall Study: More than one race | 2 | 0 | 0 | 2
  Overall Study: Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 4 | 23 | 26 | 53
  Hungary | 0 | 1 | 3 | 4
  United States | 14 | 7 | 6 | 27
  Japan | 0 | 15 | 13 | 28
  Taiwan | 0 | 3 | 7 | 10
  Poland | 0 | 3 | 1 | 4
  Australia | 0 | 5 | 2 | 7
  Spain | 0 | 7 | 5 | 12
  Singapore | 6 | 0 | 0 | 6
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: The study consists of Safety Lead-In (24 patients in Varlitinib + Capecitabine group) and Part 1 (64 patients in Varlitinib + Capecitabine group, 63 patients in Placebo + Capecitabine group)
  kg/m^2
    BMI - Safety Lead-in: number analyzed (Participants) | 24 | 0 | 0 | 24
    BMI - Safety Lead-in | 36.85 (58.381) |  |  | 36.85 (58.381)
    BMI - Part 1: number analyzed (Participants) | 0 | 64 | 63 | 127
    BMI - Part 1 |  | 24.6 (4.69) | 23.8 (4.52) | 24.2 (4.60)

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) - Part 1
Description: Part 1: The ORR was defined as the number (%) of subjects with ≥ 1 visit response of complete response (CR) or partial response (PR). Data obtained up until progression, or until last evaluable assessment in the absence of progression, was included in the assessment of ORR, regardless of whether subjects discontinued treatment or received a subsequent therapy prior to progression. Best overall RECIST Response (BOR) was calculated based on the overall visit responses from each RECIST assessment, i.e. the best response a subject had following randomization and prior to RECIST progression or the last evaluable assessment in the absence of RECIST progression. Categorization of BOR was based on the RECIST criteria using the following response categories: CR, PR, stable disease (SD), progressive disease (PD) and not evaluable (NE).
Time Frame: Data obtained up until progression, or until last evaluable assessment in the absence of progression, regardless of whether subjects discontinued treatment or received a subsequent therapy prior to progression, up to 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Varlitinib and Capecitabine | Placebo and Capecitabine
Number analyzed (Participants) | 64 | 63
Participants
  Responders - CR | 0 | 0
  Responders - PR | 6 | 3
  Non-Responders - SD | 29 | 34
  Non-Responders - PD | 24 | 24
  Non-Responders - NE | 5 | 2

2. Primary Outcome: Progression-free Survival (PFS) - Part 1
Description: Part 1: Progression-free survival (PFS) was defined as the time from randomization (or starting treatment for the Safety Lead-in) until the date of objective disease progression or death (by any cause in the absence of disease progression) regardless of whether the subject withdrew from randomized therapy or received another antitumor therapy prior to disease progression. Subjects who did not experience disease progression or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST assessment. However, if the patient progressed or died after ≥ 2 missed visits (12 weeks ± 5 days maximum), the subject was censored at the time of the latest evaluable RECIST assessment. The PFS time was based on the scan/assessment dates rather than visit dates.
Time Frame: Time from randomization until date of objective disease progression or death (by any cause in absence of disease progression) regardless of whether subject withdrew from randomized therapy or received another antitumor therapy prior to PD, up to 2 years.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Varlitinib and Capecitabine | Placebo and Capecitabine
Number analyzed (Participants) | 49 | 47
Months | 2.83 [1.48 to 5.62] | 2.79 [1.41 to 4.24]

3. Secondary Outcome: Object Response Rates (ORR) - Safety Lead-In
Description: The ORR rate was defined as the number (%) of subjects with ≥ 1 visit response of complete response (CR) or partial response (PR). Data obtained up until progression, or until last evaluable assessment in the absence of progression, was included in the assessment of ORR, regardless of whether subjects discontinued treatment or received a subsequent therapy prior to progression. In all study parts, the primary assessment of ORR was based on the Full Analysis Set (FAS).
Time Frame: Data obtained up until progression, or until last evaluable assessment in absence of progression, regardless of whether subjects discontinued treatment or received a subsequent therapy prior to progression, up to 2 years.
Measure: Count of Participants; unit: Participants
Groups:
- Varlitinib + Capecitabine: This part of the study was a single arm, open-label design to assess the safety of varlitinib (300 mg administered BID every day) plus capecitabine (1000 mg/m2 administered BID every day for 14 days, followed by a 7-day rest period) in a small set of subjects (12 to 20 subjects) with 12 subjects completing the PK and ECG evaluations. Treatment was continued until disease progression, development of unacceptable toxicity, withdrawal of consent, or death.
Arm/Group | Varlitinib + Capecitabine
Number analyzed (Participants) | 24
Participants
  Responders - CR | 0
  Responders - PR | 1
  Non-Responders - SD | 5
  Non-Responders - PD | 9
  Non-Responders - NE | 9

4. Secondary Outcome: Overall Survival (OS) - Part 1
Description: Part 1: Overall survival (OS) was defined as the time from the date of randomization until death due to any cause. Any subject not known to have died at the time of the data cut-off was censored based on the last recorded date on which the subject was known to be alive.
Time Frame: Time from the date of randomization until death due to any cause, up to 2 years
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Varlitinib and Capecitabine | Placebo and Capecitabine
Number analyzed (Participants) | 35 | 35
Months | 7.8 [4.5 to 11.5] | 7.5 [5.3 to NA] — The 75th percentile is Not Evaluable (NE), because the 75th percentile has not been reached yet (i.e. the data are too immature for that arm)

5. Secondary Outcome: Overall Survival (OS) - Safety Lead-In
Description: as for outcome 4
Time Frame: Time from the date of randomization until death due to any cause, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Varlitinib + Capecitabine
Number analyzed (Participants) | 24
Participants
  Alive | 17
  Withdrew Consent | 2
  Dead | 4
  Withdrew due to AE | 1

6. Secondary Outcome: Duration of Response (DoR) - Part 1
Description: Part 1: Duration of response (DoR) was defined as the time from the date of first documented response until the date of documented PD or death in the absence of disease progression. The end of the response should have coincided with the date of disease progression or death from any cause used for the PFS endpoint.
  For Part 1, DoR was calculated based on data from the ICR of radiological data.
Time Frame: Time from the date of first documented response until the date of documented PD or death in the absence of disease progression, up to 2 years
Population: Kaplan Meier median is presented for DoR. At the time of reporting, there were 3 censored observations in the V+C arm, none in the P+C arm. The observed number of responders in the trial was much lower than anticipated; 9 responders in total, 6 for varlitinib and 3 for placebo. Based on results of the primary endpoints, the follow-up analysis to provide more long-term efficacy data planned for when 70% of patients had experienced an OS event was not undertaken based on pre-specified criteria.
Measure: Median (Full Range); unit: Days
Arm/Group | Varlitinib and Capecitabine | Placebo and Capecitabine
Number analyzed (Participants) | 6 | 3
Days | 158 [43 to 158] | 90 [48 to 246]

7. Secondary Outcome: Disease Control Rate DCR - Part 1
Description: Part 1: DCR rate was defined as the number (%) of subjects with ≥ 1 visit response of CR or PR, or with SD for a minimum of 12 weeks (± 5 days) from randomization. Data obtained up until progression, or until last evaluable assessment in the absence of progression, were included in the assessment of DCR, regardless of whether subjects discontinued treatment or received a subsequent therapy prior to progression. For all study parts, the primary assessment of DCR was based on the FAS.
  For Part 1, DCR was calculated based on data from the ICR
Time Frame: Number (%) of subjects with ≥ 1 visit response of CR or PR, or with SD for a minimum of 12 weeks (± 5 days) from randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Varlitinib and Capecitabine | Placebo and Capecitabine
Number analyzed (Participants) | 64 | 63
Participants
  Disease Control - CR | 0 | 0
  Disease Control - PR | 6 | 3
  Disease Control - SD for 12 weeks | 12 | 16
  No Disease Control - SD < 12 weeks | 17 | 18
  No Disease Control - PD | 24 | 24
  No Disease Control - NE | 5 | 2

8. Secondary Outcome: Tumor Size - Part 1
Description: Part 1: The percentage change from baseline in tumor size at Week 12 (%ΔTSWk12) was a secondary endpoint for Part 1 and was used to present waterfall plots of the target lesion data in the Evaluable for Response (EFR) Population
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: Percentage change from Baseline
Arm/Group | Varlitinib and Capecitabine | Placebo and Capecitabine
Number analyzed (Participants) | 51 | 51
Percentage change from Baseline | 18.1 (39.46) | 22.6 (36.11)

9. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Tests- Safety Lead-in
Description: Clinical laboratory tests (hematology, clinical chemistry, urinalysis) - Number of Participants with Clinically Significant Laboratory Tests.
Time Frame: Subject screening visit to 28 days post last study drug administration
Population: No subjects reported with any CS values across majority of the hematologic, clinical chemistry, urinalysis parameters during the Safety Lead-In of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Varlitinib + Capecitabine
Number analyzed (Participants) | 24
Participants | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Tests - Part 1
Description: as for outcome 9
Time Frame: Subject screening visit to 28 days post last study drug administration
Population: No subjects reported with any CS values across majority of the hematologic, clinical chemistry and urinalysis parameters at the end of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Varlitinib and Capecitabine | Placebo and Capecitabine
Number analyzed (Participants) | 64 | 63
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Change in Vital Signs and Physical Examinations - Safety Lead-In
Description: Number of participants with clinically significant change in vital signs (blood pressure [diastolic and systolic], heart rate, respiratory rate, body temperature) and physical examination.
Time Frame: Subject screening visit to 28 days post last study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Varlitinib + Capecitabine
Number analyzed (Participants) | 24
Participants | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Change in Vital Signs and Physical Examinations - Part 1
Description: as for outcome 11
Time Frame: Subject screening visit to 28 days post last study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Varlitinib and Capecitabine | Placebo and Capecitabine
Number analyzed (Participants) | 64 | 63
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With ECG Parameters of Interest - Safety Lead-In
Description: Number of participants with ECG parameters of interest: Max. on-treatment QTcF Value: >450 to 480 msec, max. on-treatment QTcF Value: >480 to 500 msec, max. on-treatment QTcF Value: >500 msec, max. on-treatment QTcB Value: >450 to 480 msec, max. on-treatment QTcB Value: >480 to 500 msec, max. on-treatment QTcB Value: >500 msec, max. QTcF CFB Value: >30 to 60 msec, max. QTcF CFB Value: >60 msec, max. QTcB CFB Value: >30 to 60 msec, max. QTcB CFB Value: >60 msec.
Time Frame: Subject screening visit to 28 days post last study drug administration
Measure: Number; unit: participants
Arm/Group | Varlitinib + Capecitabine
Number analyzed (Participants) | 24
participants
  Maximum on-treatment QTcF Value: >450 to 480 msec | 8
  Maximum on-treatment QTcF Value: >480 to 500 msec | 0
  Maximum on-treatment QTcF Value: >500 msec | 0
  Maximum on-treatment QTcB Value: >450 to 480 msec | 10
  Maximum on-treatment QTcB Value: >480 to 500 msec | 2
  Maximum on-treatment QTcB Value: >500 msec | 0
  Maximum QTcF CFB Value: >30 to 60 msec | 8
  Maximum QTcF CFB Value: >60 msec | 1
  Maximum QTcB CFB Value: >30 to 60 msec | 6
  Maximum QTcB CFB Value: >60 msec | 1

14. Secondary Outcome: Number of Participants With ECG Parameters of Interest - Part 1
Description: Number of participants with ECG parameters of interest: Max. on-treatment QTcF Value: <=450 msec, max. on-treatment QTcF Value: >450 to 480 msec, max. on-treatment QTcF Value: >480 to 500 msec, max. on-treatment QTcF Value: >500 msec, max. on-treatment QTcB Value: <=450 msec, max. on-treatment QTcB Value: >450 to 480 msec, max. on-treatment QTcB Value: >480 to 500 msec, max. on-treatment QTcB Value: >500 msec, max. QTcF CFB Value: <=30 msec, max. QTcF CFB Value: >30 to 60 msec, max. QTcF CFB Value: >60 msec, max. QTcB CFB Value: <=30 msec, max. QTcB CFB Value: >30 to 60 msec, max. QTcB CFB Value: >60 msec.
Time Frame: Subject screening visit to 28 days post last study drug administration
Measure: Number; unit: Participants
Arm/Group | Varlitinib and Capecitabine | Placebo and Capecitabine
Number analyzed (Participants) | 64 | 63
Participants
  Maximum on-treatment QTcF Value: <=450 msec | 53 | 57
  Maximum on-treatment QTcF Value: >450 to 480 msec | 10 | 6
  Maximum on-treatment QTcF Value: >480 to 500 msec | 0 | 0
  Maximum on-treatment QTcF Value: >500 msec | 1 | 0
  Maximum on-treatment QTcB Value: <=450 msec | 42 | 40
  Maximum on-treatment QTcB Value: >450 to 480 msec | 21 | 22
  Maximum on-treatment QTcB Value: >480 to 500 msec | 0 | 1
  Maximum on-treatment QTcB Value: >500 msec | 1 | 0
  Maximum QTcF CFB Value: <=30 msec | 56 | 57
  Maximum QTcF CFB Value: >30 to 60 msec | 7 | 4
  Maximum QTcF CFB Value: >60 msec | 0 | 1
  Maximum QTcB CFB Value: <=30 msec | 55 | 54
  Maximum QTcB CFB Value: >30 to 60 msec | 8 | 7
  Maximum QTcB CFB Value: >60 msec | 0 | 1

15. Secondary Outcome: ECOG Performance Status - Part 1
Description: Eastern Cooperative Oncology Group (ECOG) Performance was clinically graded based on the following:
  Grade 0 = Normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  Grade 1 = Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Grade 2 = In bed < 50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Grade 3 = In bed > 50% of the time. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  Grade 4 = 100% bedridden. Completely disabled. Cannot carry on any self- care. Totally confined to bed or chair.
  Grade 5 = Death
Time Frame: Subject screening visit to 28 days post last study drug administration
Population: For the Varlitinib 300 mg BID + Capecitabine treatment group, ECOG Performance Status scores ranged from 0 to 3 at EOT.
  For the Placebo + Capecitabine treatment group, ECOG Performance Status scores ranged from 0 to 3 at EOT.
Measure: Count of Participants; unit: Participants
Arm/Group | Varlitinib and Capecitabine | Placebo and Capecitabine
Number analyzed (Participants) | 64 | 63
Participants
  Baseline Value Grade 0 - EOT Value Grade 0 | 16 | 11
  Baseline Value Grade 0 - EOT Value Grade 1 | 13 | 10
  Baseline Value Grade 0 - EOT Value Grade 2 | 0 | 2
  Baseline Value Grade 0 - EOT Value Grade 3 | 4 | 1
  Baseline Value Grade 0 - EOT Value Not done | 4 | 2
  Baseline Value Grade 1 - EOT Value Grade 0 | 1 | 5
  Baseline Value Grade 1 - EOT Value Grade 1 | 10 | 25
  Baseline Value Grade 1 - EOT Value Grade 2 | 5 | 2
  Baseline Value Grade 1 - EOT Value Grade 3 | 0 | 0
  Baseline Value Grade 1 - EOT Value Not done | 11 | 5

ADVERSE EVENTS:
Time Frame: Subject screening visit to 28 days post last study drug administration, up to 2 years.
Arm/Group | Varlitinib and Capecitabine - Safety Lead-In | Varlitinib and Capecitabine - Part 1 | Placebo and Capecitabine - Part 1
All-Cause Mortality (participants affected / at risk) | 2/24 | 35/64 | 35/63
Serious Adverse Events (participants affected / at risk) | 13/24 | 25/64 | 27/63
Other Adverse Events (participants affected / at risk) | 24/24 | 64/64 | 59/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varlitinib and Capecitabine - Safety Lead-In (N=24) | Varlitinib and Capecitabine - Part 1 (N=64) | Placebo and Capecitabine - Part 1 (N=63)
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 1
Bile duct obstruction (Hepatobiliary disorders) | 2 | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 4 | 4
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 4 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Lung Infection (Infections and infestations) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 3 | 0
Rash generalized (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Toxic leukoencephalopathy (Nervous system disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4 | 2
Blood bilirubin increased (Investigations) | 0 | 5 | 5
Disease progression (General disorders) | 0 | 2 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Hepatobiliary infection (Infections and infestations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hemobilia (Hepatobiliary disorders) | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 1
Embolism (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 1
Biliary sepsis (Hepatobiliary disorders) | 0 | 1 | 0
Blood culture positive (Blood and lymphatic system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Dyspnoea (Nervous system disorders) | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Hernia (Renal and urinary disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Biloma (Hepatobiliary disorders) | 0 | 1 | 0
Cholangiolitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varlitinib and Capecitabine - Safety Lead-In (N=24) | Varlitinib and Capecitabine - Part 1 (N=64) | Placebo and Capecitabine - Part 1 (N=63)
Nausea (Gastrointestinal disorders) | 15 (29) | 33 (58) | 14 (19)
Diarrhoea (Gastrointestinal disorders) | 13 (31) | 26 (43) | 16 (19)
Vomiting (Gastrointestinal disorders) | 11 (27) | 22 (30) | 11 (18)
Abdominal Pain (Gastrointestinal disorders) | 9 (12) | 16 (27) | 12 (20)
Constipation (Gastrointestinal disorders) | 8 (19) | 9 (9) | 9 (9)
Stomatitis (Gastrointestinal disorders) | 6 (9) | 7 (8) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 5 (8) | 7 (9) | 4 (4)
Ascites (Gastrointestinal disorders) | 4 (4) | 3 (3) | 4 (4)
Abdominal Distension (Gastrointestinal disorders) | 7 (13) | 4 (5) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 3 (4) | 2 (2)
Fatigue (General disorders) | 14 (35) | 16 (33) | 12 (17)
Pyrexia (General disorders) | 10 (18) | 15 (23) | 11 (13)
Asthenia (General disorders) | 5 (9) | 11 (20) | 7 (9)
Malaise (General disorders) | 2 (2) | 8 (14) | 4 (4)
Chills (General disorders) | 5 (7) | 6 (7) | 2 (2)
Mucosal Inflammation (General disorders) | 0 (0) | 5 (8) | 2 (2)
Oedema Peripheral (General disorders) | 7 (12) | 4 (5) | 3 (3)
Blood Bilirubin Increased (Investigations) | 8 (17) | 28 (71) | 14 (30)
Blood Creatinine Increased (Investigations) | 3 (5) | 15 (26) | 3 (3)
Aspartate Aminotransferase Increased (Investigations) | 5 (10) | 9 (19) | 7 (11)
Platelet Count Decreased (Investigations) | 4 (16) | 8 (13) | 8 (11)
Alanine Aminotransferase Increased (Investigations) | 4 (7) | 10 (22) | 5 (8)
Neutrophil Count Decreased (Investigations) | 2 (5) | 3 (7) | 5 (21)
Weight Decreased (Investigations) | 3 (4) | 3 (3) | 1 (1)
Palmar-plantar Erythrodysaethesia Syndrome (Skin and subcutaneous tissue disorders) | 6 (18) | 20 (32) | 19 (37)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (13) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 4 (7) | 8 (10) | 4 (7)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 12 (33) | 25 (49) | 11 (15)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 6 (11) | 5 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (20) | 2 (6) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (10) | 4 (5) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 6 (11) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 13 (30) | 14 (27)
Pneumonia (Infections and infestations) | 0 (0) | 5 (5) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (2) | 5 (8) | 2 (2)
Dizziness (Nervous system disorders) | 7 (11) | 4 (5) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (4) | 5 (6) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (16) | 5 (5) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4) | 3 (3)
Cholangitis (Hepatobiliary disorders) | 2 (5) | 5 (10) | 5 (8)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (8) | 7 (16) | 1 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (5) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (4) | 3 (4) | 3 (3)
Acute Kidney Injury (Renal and urinary disorders) | 2 (9) | 5 (6) | 1 (1)
Proteinuria (Renal and urinary disorders) | 5 (6) | 3 (6) | 2 (2)
Hypotension (Vascular disorders) | 6 (8) | 4 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (8) | 0 (0) | 1 (1)
Faeces discolored (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 2 (5) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Early satiety (General disorders) | 2 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (3) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 2 (3) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (2) | 4 (4)
International normalised ratio increased (Investigations) | 2 (3) | 1 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 2 (8) | 2 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT03093870/Prot_002.pdf
  • Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT03093870/SAP_003.pdf